CLINICAL TRIAL: NCT01838499
Title: A Phase IIa Randomized, Double-Blind, Placebo-controlled, Multicenter Study to Assess the Safety, Tolerability and Preliminary Efficacy of MEDI8968 in Subjects With Moderate to Severe Hidradenitis Suppurativa
Brief Title: Assessment of the Safety, Tolerability and Efficacy of MEDI8968 in Subjects With Moderate to Severe Hidradenitis Suppurativa
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: At the planned IA for decision making, no evidence was demonstrated of MEDI8968 activity in reducing (HS) severity or pain over that seen with placebo.
Sponsor: AstraZeneca (Industry)
Collaborators: ICON plc (Industry); Covance (Industry); PHT Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5440C00001
Record Dates: First submitted 2013-04-19; First posted 2013-04-24 (Estimated); Results first posted 2016-09-01 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-07

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MEDI8968 (Experimental)
  Interventions: Biological: MEDI8968
- Saline (Placebo Comparator)
  Interventions: Biological: Saline

INTERVENTIONS:
Biological: MEDI8968 — SC injection at baseline, Week 4 and Week 8
  Other Names: Investigational Product
  Arms: MEDI8968
Biological: Saline — SC injection at baseline, Week 4 and Week 8
  Other Names: Placebo
  Arms: Saline

SUMMARY:
The purpose of this study is to gain initial evidence for the safety, tolerability and efficacy of MEDI8968 for the treatment of subjects with moderate to severe hidradenitis suppurativa

ELIGIBILITY:
Inclusion Criteria:

* Hidradenitis suppurativa (HS) (moderate to severe)
* Diagnosis of HS for at least 1 year
* At least 5 active inflammatory lesions in at least 2 locations
* On a stable dose of antibiotics and/or analgesics for at least 4 weeks (if already taking these medications)
* Average pain score of 3-9.

Exclusion Criteria:

* History of cyclic neutropenia
* Laboratory assessment abnormalities
* Underlying disorder considered unsuitable for inclusion
* Other skin diseases that may interfere with HS assessment
* Pregnancy or planning for pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2013-05; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert AK Lee, MD, Principal Investigator — University of California, San Diego
Locations (27):
- United States (27):
  - Research Site, Phoenix, Arizona
  - Research Site, Bakersfield, California
  - Research Site, Fremont, California
  - Research Site, Los Angeles, California
  - Research Site, San Diego, California
  - Research Site, San Francisco, California
  - Research Site, Miami, Florida
  - Research Site, Orange Park, Florida
  - Research Site, Ormond Beach, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Macon, Georgia
  - Research Site, Skokie, Illinois
  - Research Site, West Dundee, Illinois
  - Research Site, Evansville, Indiana
  - Research Site, Indianapolis, Indiana
  - Research Site, Rockville, Maryland
  - Research Site, St Louis, Missouri
  - Research Site, Forest Hills, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, High Point, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Hershey, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Rapid City, South Dakota
  - Research Site, Arlington, Texas
  - Research Site, Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 221 subjects enrolled, 109 randomised. Enrolment for ERF based on info databased, as per programmed outputs and the CSR - the criteria being to have provided written consent. 3 additional patients were accounted for in the PRF. M and F subjects with moderate to severe HS were randomised to MEDI8968 or Placebo. 29 centres in the US involved.
Pre-assignment Details: Randomisation to treatment was stratified by PGA score on the day of randomisation (Stratum 1=PGA score of 3; Stratum 2=PGA score of 4 or 5).
Groups:
- MEDI8968; Saline: SC injection
Period: Overall Study
Arm/Group | MEDI8968 | Saline
Started | 55 | 54
Completed | 31 | 37
Not Completed | 24 | 17
Not completed — Protocol Violation | 0 | 1
Not completed — Lost to Follow-up | 2 | 4
Not completed — Lack of Efficacy | 1 | 2
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 19 | 9

BASELINE CHARACTERISTICS:
Population: Full Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | MEDI8968 | Saline | Total
Number analyzed (Participants) | 55 | 54 | 109
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.5 (11.08) | 36.4 (12.42) | 36.9 (11.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 38 | 83
  Male | 10 | 16 | 26

OUTCOME MEASURES:

1. Primary Outcome: 1) Percentage of Subjects Achieving a Clinically Relevant Response in Physician Global Assessment (PGA), With Score 0,1 or 2 From Baseline to 12 Weeks
Description: Percentage of subjects achieving a clinically significant response measured by the proportion of subjects who achieve 0, 1, or 2 PGA by the end of week 12
Time Frame: 12 weeks
Population: FAS
Measure: Number; unit: % of patients
Arm/Group | MEDI8968 | Saline
Number analyzed (Participants) | 55 | 54
% of patients
  Responders (%) | 23.6 | 18.5
  Non-responders (%) | 76.4 | 81.5
Statistical Analysis 1: Comparison: MEDI8968 vs Saline; Analysis of proportion of Responders for Physician's Global Assessment (PGA score 0, 1 or 2) at Week 12 - LOCF. Difference in proportions MEDI8968 - placebo. Wald asymptotic confidence limits calculated; Test type: Superiority or Other; p > 0.05, Mixed Models Analysis; Difference in proportions = 0.051, 80% CI 2-sided [-0.067 to 0.169] — MEDI8968 - placebo

2. Secondary Outcome: 2) Subject's Global Impression of Change Reported on PGIC Scale (1-7 Point Scale Ranging From 1 "Very Much Improved" to 7 "Very Much Worse")
Description: Percentage of subjects achieving a clinically significant response measured by the proportion of subjects who are "minimally improved", "much improved" or "very much improved" on the Patient's Global Impression of Change (PGIC)
Time Frame: 12 weeks
Measure: Number; unit: % of patients
Arm/Group | MEDI8968 | Saline
Number analyzed (Participants) | 55 | 54
% of patients
  Responders (%) | 49.1 | 55.6
  Non-Responders (%) | 50.9 | 44.4
Statistical Analysis 1: Comparison: MEDI8968 vs Saline; Difference in proportions MEDI8968 - placebo. Wald asymptotic confidence limits calculated; Test type: Superiority or Other; p > 0.05, Mixed Models Analysis; Difference in proportions = -0.065, 80% CI 2-sided [-0.205 to 0.076]

3. Secondary Outcome: Change From Baseline to 12 Weeks in Numerical Assessment Scale Numerical Rating Scale for Pain
Description: Assessment of change in pain via Numerical Rating Scale. Daily pain is reported by the subject using an 11-point 0 (no pain) to 10 (worst pain imaginable) numeric rating scale.
  Baseline score is the average of the values collected in the 7 days prior to first dose of study drug. Each Visit score is the average of the values collected in the 7 days prior to that visit.
Time Frame: 12 weeks
Population: FAS (LOCF)
Measure: Least Squares Mean (Standard Error); unit: changes in scores on a scale
Arm/Group | MEDI8968 | Saline
Number analyzed (Participants) | 50 | 50
changes in scores on a scale
  Week 4 | -1.09 (0.35) | -1.02 (0.36)
  Week 8 | -1.76 (0.36) | -1.31 (0.36)
  Week 12 | -1.79 (0.46) | -1.76 (0.47)
Statistical Analysis 1: Comparison: MEDI8968 vs Saline; Analysis of change from baseline (Week 12) estimated from ANCOVA model with tmt group and PGA stratum at randomisation included in the model and average daily pain at baseline as a covariate; Test type: Superiority or Other; p = 0.945, ANCOVA; Change from baseline (at week 12) = -0.03, 80% CI 2-sided [-0.63 to 0.57] — MEDI8968 - Placebo

ADVERSE EVENTS:
Time Frame: 24 weeks. However, if a subject withdraws from treatment for any reason prior to week 24, the subject should continue to be seen up to 16 weeks after his/her last dose.
Description: In the tables below all the SAEs are presented. In the Other Adverse events tables please note that a Frequency Threshold of 5% has been applies to reporting the AEs and associated summaries. If, within a treatment group the frequency >= 5%, the associated information has been presented for both treatment arms.
Arm/Group | MEDI8968 | Saline
Serious Adverse Events (participants affected / at risk) | 2/55 | 2/54
Other Adverse Events (participants affected / at risk) | 8/55 | 2/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI8968 (N=55) | Saline (N=54)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pheumonia (Infections and infestations) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI8968 (N=55) | Saline (N=54)
Pheumonia (Infections and infestations) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Fatigue (General disorders) | 3 (3) | 0 (0)

LIMITATIONS AND CAVEATS:
The trial terminated early due to lack of efficacy. An interim analysis was conducted after the first 61 subjects at 12 weeks and showed no evidence of MEDI8968 activity in reducing (HS) severity or pain over that seen with placebo.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No